CLINICAL TRIAL: NCT02221635
Title: A Study to Evaluate the Efficacy of Repetitive Transcranial Magnetic Stimulation in the Prevention of Relapse of the Symptoms of Schizoaffective Disorder
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation in the Prevention of Relapse of Schizoaffective
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: The No.3 hospital of PLA (Unknown); The No.91 hospital of PLA (Unknown); No. 102 Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Sponsor
Other Study IDs: Yunchun Chen; Xijing H (Registry Identifier: XijingH)
Record Dates: First submitted 2012-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Schizoaffective Disorder
Keywords: Schizoaffective Disorder; Repetitive transcranial magnetic stimulation (rTMS)
MeSH Terms: conditions — Psychotic Disorders | interventions — Transcranial Magnetic Stimulation; Risperidone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- rTMS+Risperidone: Intensity of 120% of individually determined motor threshold; frequency : 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s.5 sessions per week for 4-6 weeks,than 2 sessions per week for 2 months, repeat that for 12 months.At the same time,risperidone (2-4mg) was took orally.
  Interventions: Procedure: rTMS + risperidone
- Risperidone: Risperidone (2-4mg) was took orally.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Procedure: rTMS + risperidone — Intensity of 120% of individually determined motor threshold; frequency : 1 Hz; 360 impulsions; on period : 1 min; off period : 30 s.5 sessions per week for 4-6 weeks,than 2 sessions per week for 2 months, repeat that for 12 months. Meanwhile,risperidone (2-4 mg) was took orally.
  Groups: rTMS+Risperidone
Drug: Risperidone — Risperidone (2-4 mg) was took orally.
  Groups: Risperidone

SUMMARY:
The purpose of this study is to evaluate the efficacy of repetitive transcranial magnetic stimulation in the prevention of relapse of the symptoms of schizoaffective disorder. Primary Outcome Measures:Time between subject randomization to treatment and the first occurrence of a relapse during the Relapse Prevention Period. Secondary Outcome Measures: Symptom change as measured by the Positive and Negative Syndrome Scale (PANSS) total and PANSS factor scores; Illness severity change as measured by Clinical Global Impression of Severity for depression (CGI-S-DEP); Change in subject functioning using the Personal and Social Performance Scale; Change in subject medication satisfaction using the Medication Satisfaction Questionnaire (MSQ).

DETAILED DESCRIPTION:
Schizoaffective disorder is a chronic illness and generally requires life-long treatment. To date however, no physical therapy has been evaluated in the maintenance treatment of schizoaffective disorder. This is a randomized (study drug assigned by chance), double-blind (neither physician nor patient knows the name of the assigned drug), medication-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of repetitive transcranial magnetic stimulation(rTMS), as monotherapy or as an adjunct to antipsychotic, relative to antipsychotic drugs in delaying the time to relapse in patients with schizoaffective disorder. Patients with acute symptoms of schizoaffective disorder will be enrolled. The study will consist of 4 periods: an up to 7 days screening/tolerability period, a 6-week open-label flexible dose lead-in period, a 6-week open-label fixed dose stabilization period, and a 12 months double-blind relapse prevention period. Patients without previous exposure to rTMS will be given 4 to 6 days of rTMS for tolerability testing. Patients can continue their current antipsychotic drugs through Day-1 (the day before the start of the study period). During the open-label periods, all patients will be treated with Risperidone. Patients who meet pre-determined stabilization criteria will be eligible to enter the double-blind relapse prevention period and will be randomly assigned to either receive rTMS or rTMS+Risperidone treatment. Efficacy will be evaluated during the study using a relapse assessment(time between subject randomization to treatment and the first occurrence of a relapse during the Relapse Prevention Period). Secondary Outcome Measures:Secondary Outcome Measures: Symptom change as measured by the Positive and Negative Syndrome Scale (PANSS) total and PANSS factor scores; Illness severity change as measured by Clinical Global Impression of Severity for depression(CGI-S-DEP); Change in subject functioning using the Personal and Social Performance Scale; Change in subject medication satisfaction using the Medication Satisfaction Questionnaire (MSQ). Safety will be assessed throughout the study by monitoring of adverse events, clinical laboratory tests, electrocardiograms (ECGs), vital sign measurements (temperature, pulse, and blood pressure), and weight. A 10 milliliter pharmacogenomic blood sample (sample for DNA research) will be collected from patients who give separate written informed consent for this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV (Diagnostic and Statistical Manual of Mental Disorders-IV)diagnosis of schizoaffective disorder
* Experiencing an acute exacerbation of psychotic symptoms
* A score of >=4 on at least 3 of the following 7 PANSS items: Delusions (P1), Hallucinatory behavior (P3), Excitement (P4), Hostility (P7), Tension (G4), Uncooperativeness (G8), and Poor Impulse Control (G14)
* A score of >=16 on YMRS and/or a score of >=16 on the HAM-D-21
* Healthy based on physical examinations, electrocardiogram (ECG), laboratory tests, medical history, and vital signs measurements

Exclusion Criteria:

* A primary active mental illness diagnosis other than schizoaffective disorder
* Have attempted suicide within 12 months or are at imminent risk of suicide or violent behavior
* Subjects with first episode of psychosis
* Received electroconvulsive therapy in the past 3 months
* History of hypersensitivity to or intolerance of paliperidone, risperidone, or 20% Intralipid (placebo)
* Received long-acting antipsychotic medication within 2 injection cycles
* Received therapy with clozapine within 3 months
* A history of neuroleptic malignant syndrome
* Previous history of lack of response to antipsychotic medication
* Subjects receiving therapy with antidepressants or mood stabilizers that has been initiated and/or changed in dose <30 days prior to screening
* Receiving therapy with carbamazepine
* Receiving therapy with monoamine oxidase inhibitors
* Pregnant, breast-feeding, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages Eligible for Study: 18 Years to 65 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: No
Sampling Method: Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Time for relapse | Monthly during the 15 month double-blind Relapse Prevention Period.
  Time between subject randomization to treatment and the first occurrence of a relapse during the Relapse Prevention Period.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | Up to 15 Months
  Symptom change as measured by the Positive and Negative Syndrome Scale (PANSS) total and PANSS factor scores
Clinical Global Impression of Severity for Schizoaffective Disorder | Up to 15 Months
  Illness severity change as measured by Clinical Global Impression of Severity for Schizoaffective Disorder (CGI-S-SCA)
Personal and Social Performance Scale | Up to 15 Months
  Change in subject functioning using the Personal and Social Performance Scale (PSP)
Change in mood symptoms | Up to 15 Months
  Change in mood symptoms as measured by YMRS (Young Mania Rating Scale,in subjects with YMRS=16 at enrollment) and HAM-D-21) (in subjects with HAM-D-21=16 at enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Tan QingRong, MD, Study Chair — XiJing Hospital, Xi'An, Shanxi, China
Locations (1):
- Qingrong, Xi'an, Shaanxi, China